CLINICAL TRIAL: NCT02160002
Title: Incubator Weaning of Moderately Preterm Infants: A Randomized Controlled Trial
Brief Title: Incubator Weaning of Moderately Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0054
Record Dates: First submitted 2014-05-08; First posted 2014-06-10 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Moderate Preterm
Keywords: Incubator Weaning; Moderately Preterm Infants; Growth Velocity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lower Weight (1600 grams) (Active Comparator): Weaning from an incubator at a lower weight (1600 grams)
  Interventions: Procedure: Weaning from an incubator at a lower weight (1600 grams)
- Higher Weight (1800 grams) (Active Comparator): Weaning from an incubator at a higher weight (1800 grams)
  Interventions: Procedure: Weaning from an incubator at a higher weight (1800 grams)

INTERVENTIONS:
Procedure: Weaning from an incubator at a lower weight (1600 grams) — Infants will be weaned from an incubator at a lower weight (1600 grams)
  Arms: Lower Weight (1600 grams)
Procedure: Weaning from an incubator at a higher weight (1800 grams) — Infants will be weaned from an incubator at a higher weight (1800 grams)
  Arms: Higher Weight (1800 grams)

SUMMARY:
The objective of this proposal is to evaluate whether weaning from an incubator to a crib at lower versus higher weight, 1600g or 1800g will result in shorter length of hospital stay among moderately preterm infants.

The hypothesis of this study is that length of hospital stay (from birth to discharge) will be decreased among moderate preterm infants weaned from an incubator to an open crib at a lower versus higher weight, 1600g vs. 1800g.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 29 0/7 to 33 6/7 weeks at birth
* Birth weight less than 1600 grams
* Greater than 48 hours of age
* Current weight less than 1540 grams
* In an incubator

Exclusion Criteria:

* Receiving phototherapy
* Receiving respiratory support (including CPAP, ventilation, HFNC > 2 LPM)
* Receiving blood pressure support
* Designated for transfer to referral hospital while in incubator
* Known major congenital or chromosomal anomaly

Ages: 29 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 366 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele C Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Seetha Shankaran, MD, Study Chair — Wayne State University; David Carlton, MD, Principal Investigator — Emory University; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Brenda B Poindexter, MD, Principal Investigator — Indiana University; Abbot Laptook, MD, Principal Investigator — Brown University, Women & Infants Hosptial of Rhode Island; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Kathleen A Kennedy, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Mike Cotten, MD, Principal Investigator — Duke University; Edward F Bell, MD, Principal Investigator — University of Iowa; Kristi Watterberg, MD, Principal Investigator — University of New Mexico; Barbara Schmidt, MD, Principal Investigator — University of Pennsylvania; Carl T D'Angio, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Pablo Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Abhik Das, PhD, Principal Investigator — RTI International
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Chowdhary V, Shukla A. Weaning of moderately preterm infants from the incubator to the crib: a randomized clinical trial. Acta Paediatr. 2019 Jul;108(7):1364. doi: 10.1111/apa.14774. Epub 2019 Apr 29. No abstract available. PMID 31033050
- [Derived] Shankaran S, Bell EF, Laptook AR, Saha S, Newman NS, Kazzi SNJ, Barks J, Stoll BJ, Bara R, Gabrio J, Childs K, Das A, Higgins RD, Carlo WA, Sanchez PJ, Carlton DP, Pavageau L, Malcolm WF, D'Angio CT, Ohls RK, Poindexter BB, Sokol GM, Van Meurs KP, Colaizy TT, Khmour A, Puopolo KM, Garg M, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health, and Human Development Neonatal Research Network. Weaning of Moderately Preterm Infants from the Incubator to the Crib: A Randomized Clinical Trial. J Pediatr. 2019 Jan;204:96-102.e4. doi: 10.1016/j.jpeds.2018.08.079. Epub 2018 Oct 15. PMID 30337189
- See also: NICHD Neonatal Research Network site — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — http://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/overview.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1565 infants were screened for eligibility. 1199 infants were excluded. 680 were excluded due to not meeting all eligibility conditions, 510 did not get consent for randomization, and 9 were consented but not randomized due to parent (1 infant) or doctor withdrawal (1 infant), becoming medically unstable (3 infants) or other reasons (4 infants).
Period: Overall Study
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Started | 187 | 179
Primary Outcome | 185 | 178
Completed | 185 | 178
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: A total of 366 infants were randomized in the study. 187 infants were randomized to the Lower Weight group. 179 infants were randomized to the Higher Weight group. The baseline statistics are based on the number of mothers or infants for whom data were available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams) | Total
Number analyzed (Participants) | 187 | 179 | 366
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational Age | 31.2 (1.3) | 31.1 (1.2) | 31.1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 87 | 180
  Male | 94 | 92 | 186
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 76 | 72 | 148
  White | 99 | 97 | 196
  Other | 12 | 10 | 22
Postmenstrual (PMA) age at start of weaning [Mean (Standard Deviation); unit: weeks] | 33.8 (1.3) | 34.3 (1.2) | 34.1 (1.3)
Maternal Age [Mean (Standard Deviation); unit: years] | 28.8 (5.8) | 28.9 (6.1) | 28.8 (5.9)
Cesarean Delivery [Count of Participants; unit: Participants] | 136 | 122 | 258

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay (LOS) From Birth to Discharge (up to 120 Days)
Description: Number of days the infant stays in hospital after birth until discharge home (up to 120 days).
Time Frame: From birth through discharge
Population: 185 infants in the lower weight group and 178 infants in the higher weight group have the date of discharge available.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 185 | 178
days | 43 [32 to 55] | 41 [33 to 52]

2. Secondary Outcome: Length of Stay (LOS) Following Weaning From Incubator to Crib to Hospital Discharge (up to 120 Days)
Description: Among infants who were successfully weaned, the number of days in the hospital counting from the start of weaning from the incubator to the crib through discharge from the hospital (up to 120 days).
Time Frame: From start of weaning from the incubator to crib through discharge (up to 120 days)
Population: There were 163 infants in the Lower Weight group that were successfully weaned from incubator to the crib; discharge date was missing for one of these infants. There were 159 infants in the Higher Weight group that were successfully weaned from incubator to the crib; 4 infants were missing start of weaning dates because of protocol violations.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 162 | 155
days | 24 [14 to 35] | 19 [10 to 26]

3. Secondary Outcome: Failure Rate of Weaning to Crib (Number of Infants With Axillary Temperature < 36.3°C After 2 Weaning Attempts)
Description: Failure of wean is defined as axillary temperature less than 36.3°C after one hour in the crib on 2 successive readings, 3 to 4 hours apart, within 24 hours of weaning to the crib in spite of additional clothes/coverings.
Time Frame: Through completion of 2 weaning attempts
Population: 178 infants in the Lower Weight group and 167 infants in the Higher Weight group have the data on whether weaning from incubator to crib was successful after two attempts at weaning.
Measure: Count of Participants; unit: Participants
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 178 | 167
Participants | 15 | 8

4. Secondary Outcome: Growth Velocity (Weight in Grams/kg/Day) From Start of Weaning From Incubator (Following Random Assignment) to 36 Weeks Postmenstrual Age (PMA)
Description: Growth velocity in terms of weight (g/kg/day), considering infant weight at start of weaning from incubator to crib (following random assignment) and weight at 36 weeks postmenstrual age (PMA).
Time Frame: Start of weaning from incubator through 36 weeks postmenstrual age (PMA)
Population: There were 257 (136 LW and 121 HW) infants who remained in the hospital at 36 weeks PMA that have weights measured at 36 weeks PMA. Twenty six infants (10 LW and 16 HW) who were still in the incubator at 36 weeks PMA and 20 infants (7 LW and 13 HW) missing the date of start of weaning were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: grams/kilograms/day
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 119 | 92
grams/kilograms/day | 15.8 (4.8) | 15.8 (4.1)

5. Secondary Outcome: Growth Parameters: Weight at Status
Description: Infant weight at status is measured at the time of discharge, death, transfer to another facility, or 120 days.
Time Frame: Status (discharge, death, transfer to another facility, or 120 days)
Population: 185 infants in the Lower Weight group and 177 infants in the Higher Weight group had their weights recorded upon reaching status.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 185 | 177
grams | 2336.3 (648.0) | 2353.6 (522.0)

6. Secondary Outcome: Growth Parameters: Length at Status
Description: Infant length at status is measured at the time of discharge, death, transfer to another facility, or 120 days.
Time Frame: Status (discharge, death, transfer to another facility, or 120 days)
Population: 174 infants in the Lower Weight group and 169 infants in the Higher Weight group have the length at status data.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 174 | 169
centimeters | 44.6 (3.2) | 44.9 (2.9)

7. Secondary Outcome: Growth Parameters: Head Circumference at Status
Description: Infant head circumference at status is measured at the time of discharge, death, transfer to another facility, or 120 days.
Time Frame: Status (discharge, death, transfer to another facility, or 120 days)
Population: 182 infants in the Lower Weight group and 173 infants in the Higher Weight group have the head circumference at status data.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 182 | 173
centimeters | 31.9 (2.2) | 32.0 (2.0)

8. Secondary Outcome: Postmenstrual Age (PMA) at Discharge
Description: Postmenstrual age (PMA) at discharge is the sum of the gestational age of the infant and its length of stay in hospital from birth to discharge.
Time Frame: Discharge
Population: 185 infants in the Lower Weight group and 178 infants in the Higher Weight group have postmenstrual age (PMA) at discharge data.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 185 | 178
weeks | 37.1 [36.3 to 38.9] | 37.0 [36.0 to 38.3]

9. Secondary Outcome: Readmission to the Hospital Within 1 Week of Discharge
Description: Number of infants re-hospitalized within 1 week (7 days) of discharge.
Time Frame: Discharge through 1 week after discharge.
Population: 174 infants in the Lower Weight group and 168 infants in the Higher Weight group had post discharge follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 174 | 168
Participants | 6 | 2

10. Secondary Outcome: Death Among Enrolled Infants
Time Frame: Status (discharge, death, transfer to another facility, or 120 days)
Population: 185 infants in the Lower Weight group and 178 infants in the Higher Weight group have status data.
Measure: Count of Participants; unit: Participants
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 185 | 178
Participants | 0 | 0

11. Secondary Outcome: Transferred to a Non-Network Hospital
Description: Number of infants transferred to another non-Network hospital.
Time Frame: Status (discharge, death, transfer to another facility, or 120 days)
Population: 185 infants in the Lower Weight group and 178 infants in the Higher Weight group have status data.
Measure: Count of Participants; unit: Participants
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 185 | 178
Participants | 11 | 9

12. Secondary Outcome: Length of Stay (LOS) Following Randomization to Hospital Discharge
Description: The number of days the infant stayed in hospital after randomization to the study until discharge.
Time Frame: From randomization through discharge.
Population: 185 infants in the Lower Weight group and 178 infants in the Higher Weight group have the date of discharge.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 185 | 178
days | 28 [19 to 39] | 27.5 [20 to 37]

13. Post Hoc Outcome: Growth Velocity (g/kg/Day) After Transfer to Crib From Incubator to Crib to 36 Weeks Postmenstural Age (PMA)
Description: Growth velocity in terms of weight (g/kg/day), considering infant weight at 24 hours after successful wean to crib and weight at 36 weeks postmenstrual age (PMA).
Time Frame: 24 hours after successful wean to 36 weeks postmenstrual age (PMA)
Population: 257 infants (136 LW, 121 HW) remained in hospital at 36 weeks PMA w/ weight measured at 36 weeks PMA. 26 (10 LW, 16 HW) were still in incubator at 36 weeks PMA, 31 (16 LW, 15 HW) were missing weight after 24 hrs of successful wean, and 4 (LW) w/ weights measured at 24 hrs after successful wean were missing date of 24 hr weight after successful wean
Measure: Mean (Standard Deviation); unit: grams/kilograms/day
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
Number analyzed (Participants) | 106 | 90
grams/kilograms/day | 11.0 (7.4) | 9.6 (7.0)

ADVERSE EVENTS:
Time Frame: Adverse events are monitored from the time of randomization through 72 hours post study intervention completion. The study intervention period is defined as from the time of randomization to the end of a successful wean or failure.
Description: Potential adverse events include inability to maintain temperature in crib, bradycardia, weight loss or lack of weight gain and feeding intolerance during the safety monitoring period.
Arm/Group | Lower Weight (1600 Grams) | Higher Weight (1800 Grams)
All-Cause Mortality (participants affected / at risk) | 0/187 | 0/179
Serious Adverse Events (participants affected / at risk) | 1/187 | 0/179
Other Adverse Events (participants affected / at risk) | 19/187 | 7/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Weight (1600 Grams) (N=187) | Higher Weight (1800 Grams) (N=179)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Weight (1600 Grams) (N=187) | Higher Weight (1800 Grams) (N=179)
Moderate cold stress (Metabolism and nutrition disorders) | 10 (10) | 3 (3)
Severe cold stress (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (3) | 2 (3)
Feeding Intolerance (Gastrointestinal disorders) | 1 (3) | 2 (3)
Desaturations (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NEC IIa (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia with desaturations (Cardiac disorders) | 1 (1) | 0 (0)
Increasing heart failure (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies.